CLINICAL TRIAL: NCT06470464
Title: Clinical Study of Thalidomide Combined With Chemotherapy in the Treatment of Relapsed or Refractory Yolk Sac Tumor in Children
Brief Title: Thalidomide Combined With Chemotherapy in the Treatment of Relapsed or Refractory Yolk Sac Tumor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shandong First Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HERO2022
Record Dates: First submitted 2024-06-17; First posted 2024-06-24 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2021-11

CONDITIONS: Germ Cell Tumor; Yolk Sac Tumor
Keywords: relapsed or refractory yolk sac tumor; thalidomide
MeSH Terms: conditions — Neoplasms, Germ Cell and Embryonal; Endodermal Sinus Tumor; Recurrence | interventions — 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- thalidomide combined with chemotherapy in the treatment of relapsed or refractory yolk sac tumor (Experimental): This study employed an open single-group clinical laboratory design method (Simon Phase II study) to investigate the efficacy and safety of combining thalidomide with TGA chemotherapy (nab-paclitaxel + gemcitabine+ epirubicin) in the treatment of children with recurrent or refractory YST. AFP levels were assessed after each course of treatment, while imaging evaluations were conducted every two courses. The remission rate following chemotherapy in this single-group clinical trial was compared to that reported in the literature for treating recurrent or refractory yolk sac tumor, evaluating overall remission rate (ORR) and event-free survival rate (EFS), as well as monitoring and recording chemotherapy-related side effects.
  Interventions: Drug: Thalidomide combined with TGA chemotherapy (nab-paclitaxel + gemcitabine+ epirubicin)

INTERVENTIONS:
Drug: Thalidomide combined with TGA chemotherapy (nab-paclitaxel + gemcitabine+ epirubicin) — The oral dose of thalidomide is 1.5-2.5mg/kg/d daily (maximum 28g). Each cycle lasts for 21 days (every three weeks), and if treatment parameters are met as described in the study, cycle two and subsequent cycles begin on day 22. Treatment will be discontinued if there is drug-related dose-limiting toxicity or disease progression. Tumor response assessment will be repeated using AFP and LDH every one cycle and imaging examination every two cycles. Children who complete the trial may continue this regimen or undergo surgery or radiation therapy if their disease goes into remission.

SUMMARY:
Remarkable progress has been made in treating germ-cell tumor (GCT) through the use of platinum-based regimens. However, part of yolk sac tumor (YST) with cisplatin resistance or recurrence is nevertheless prone to relapse after second-line treatment. This leaves a gap in effective treatment, which needs to be filled by novel therapeutic approaches. This paper is the first one to report the treatment combining thalidomide with nab-paclitaxel, gemcitabine, and epirubicin (T-TGA) for children with repeated relapsed or refractory yolk sac tumor (rrrYST).

DETAILED DESCRIPTION:
Thalidomide (THD) is currently widely used in the treatment of immune rheumatic diseases, blood tumors and solid tumors. Solid tumors are mostly used in the treatment of lung cancer, liver cancer, stomach cancer, colorectal cancer, pancreatic cancer, etc., and are limited to patients with advanced or advanced tumors. The main mechanisms of its action are inhibition of angiogenesis, immune regulation, induction of apoptosis, target teratogenesis and so on. However, whether from animal experiments or clinical studies, thalidomide alone or in combination with chemotherapy has not been seen to have a very effective therapeutic effect or exact clinical application in the treatment of these solid tumors.

According to the latest relevant case analysis reports and clinical trial results abroad, TIP regimen is still the priority recommended treatment regimen in the previous data for children with recurrent and refractory malignant germ cell tumors. However, the combination of Sirolimus and TIC regimen (nab-paclitaxel + isocyclophosphamide + carboplatin) previously explored by our research group can greatly improve the remission rate of recurrent and refractory germinal cell tumors, especially for recurrent and refractory yolk sac tumors, a certain proportion can be cured or the opportunity for surgery and radiotherapy can be obtained to achieve cure. However, there are still some children who are insensitive or progress again after 2 cycles of remission. For these children with multiple relapsed or particularly difficult yolk sac tumors, there is no effective treatment plan in the world at present, and there is no relevant clinical trial. However, through our clinical experience and understanding in the treatment process of these children, The results of thalidomide combined with TGA chemotherapy regimen (nab-paclitaxel + gemcitabine + epirubicin) were satisfactory. Therefore, we hope to evaluate the therapeutic effectiveness and adverse reactions of this regimen through clinical trials, so as to provide an effective treatment option for children with recurrent and refractory yolk sac tumor.

This paper is the first one to report the treatment combining thalidomide with nab-paclitaxel, gemcitabine, and epirubicin (T-TGA) for children with repeated relapsed or refractory yolk sac tumor (rrrYST).

ELIGIBILITY:
Inclusion Criteria:

1. The child must have histological evidence of an extracranial malignant germ cell tumor (vitelline sac tumor).
2. Children must be no more than 18 years old at the time of study participation.
3. The patients were children with vitelline cystic tumor who were resistant to drugs after at least two platinum-containing chemotherapy regimes or whose disease recurred within 3 months after chemotherapy regimes, or who recurred again or repeatedly after treatment with Sirolimus combined with TIC chemotherapy regimes.
4. The child must have measurable lesions (recorded according to RECIST criteria) or non-evaluable disease with tumor marker AFP greater than 5 times the upper limit of normal.
5. Lansky performance status score ≥50.
6. The life expectancy of the child must exceed 6 weeks.
7. The child must have recovered from the response to all previous anticancer treatments.
8. No serious organ dysfunction: normal cardiac function (ejection fraction > 50% or BNP < 2000pg/ml); Liver function: alanine aminotransferase increased less than 5 times the upper limit of normal, bilirubin increased less than 3 times the upper limit of normal; Renal function: creatinine and urea nitrogen levels below the normal range; The white blood cells were greater than 3×109/L, and the platelets were greater than 100×109/L.
9. Obtain the informed consent of the guardian and sign the informed consent.

Exclusion Criteria:

1. Patients with other tumors.
2. Heart, brain, liver, kidney and other organ failure patients.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2024-06-16 (Actual); Study Completion 2024-06-16 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Every 3 weeks per cycle, up to 6 cycles
  Proportion of participants achieving partial or complete response，Measurement: Imaging (CT/MRI) every 2 cycles per RECIST 1.1；Serum AFP reduction ≥90% from baseline.

SECONDARY OUTCOMES:
Radiographic Tumor Response Evaluation | Every 6 weeks (i.e., every 2 chemotherapy cycles)
  Assessment of tumor size and characteristics to evaluate treatment response. Method: Contrast-enhanced computed tomography (CT) or magnetic resonance imaging (MRI) scans Outcome Metrics: Complete response (CR), partial response (PR), stable disease (SD), or progressive disease (PD) based on RECIST 1.1 criteria

CONTACTS AND LOCATIONS:
Overall Officials: Jingfu Wang, MD, Study Director — Shandong Cancer Hospital and Institute
Locations (1):
- Shandong Cancer Hospital and Institute, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No